CLINICAL TRIAL: NCT00195195
Title: A Rapamune Follow-up Registry in Transplant Recipients in the Nordic Countries, "Wrap-up"
Brief Title: Study Evaluating Rapamune in Transplant Recipients in the Nordic Countries
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0468-101157
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Transplantation
Keywords: Transplantation
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Sirolimus
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Transplantation patients treated with sirolimus who consent to participate in the study (register)
  Other Names: Rapamune

SUMMARY:
The purpose of this study is to gather information about the long-term effects and safety of treatment with Rapamune in transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Transplantation patients treated with sirolimus (Rapamune).

Exclusion Criteria:

* Patients must be able to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Transplantation patients treated with sirolimus.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala